CLINICAL TRIAL: NCT06296901
Title: o Wipe or Not To Wipe?: That Is The Question
Brief Title: To Wipe or Not To Wipe?: That Is The Question
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna A. Orzel (Other)
Responsible Party: Sponsor-Investigator, Joanna A. Orzel, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202310353
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineal Wipe (Experimental): Patient will use wipe before collecting mid-stream clean catch culture
  Interventions: Other: Perineal Wipe
- No Wipe (No Intervention): Patient will not use wipe before collecting mid-stream clean catch culture

INTERVENTIONS:
Other: Perineal Wipe — use of perineal wipe
  Other Names: PDI Castile Soap Towelettes
  Arms: Perineal Wipe

SUMMARY:
The primary aim of this randomized control trial is to characterize whether a mid-stream clean catch sample using a cleansing wipe in the setting of symptomatic UTI in a female patient is associated with a lower rate of contamination. We hypothesize that using a perineal cleansing wipe at the time of a midstream urine sample will decrease rates of contamination for female patients with a symptomatic UTI.

DETAILED DESCRIPTION:
The primary aim of this study is to determine whether using a perineal cleansing wipe decreases the rate of a contaminated midstream clean catch sample in female patients with a symptomatic UTI.

This is a single-blind, randomized controlled trial comparing the use of a perineal cleansing wipe versus no wipe in adult female patients who present to the urology clinic at IRL or 3RC with a symptomatic UTI.

Following IRB approval, patients who are eligible for the study (female patients >18 years of age with active UTI symptoms) will be asked to participate in the study. After obtaining informed consent, participants will be randomized using a validated web-based randomization tool. Patients who are randomized to receive a wipe will receive verbal and printed/visual instructions to take with them for sample collection.

Patients who are asymptomatic, have an indwelling catheter, SPT, stent, nephrostomy tube, perform CIC, are on daily antibiotic prophylaxis, or already on existing antibiotics will be excluded.

The study will be open for approximately 1 year to enroll participants.

The following data will be collected via chart review and entered into a REDCap database: age, BMI, UTI symptoms (urgency, frequency, urgency urinary incontinence increased from baseline symptoms, dysuria, fevers, flank pain, suprapubic pain/pressure, low back pain, cloudy urine, malodorous urine), urinalysis and microscopy data (if ordered), final culture result including contamination type (multiple organisms, skin flora, urogenital flora, group B streptococcus, lactobacillus), antibiotic treatment.

Sample size calculations were performed based on an expected 60% contamination rate for the no wipe group. If an anticipated maximum contamination rate of 50% for the wipe group, that provides a 10% between-group difference. For an N=600, even allocation provides 300 patients per group. There would be 69.3% power when testing for a between-group difference at alpha = 0.05.

Demographics of the patients will be assessed via summary statistics. Comparisons between the demographics of the two groups will be made using Fisher's Exact or chi squared tests for categorical variables and using T-test or Wilcoxon rank sum tests for continuous variables, where appropriate. Primary outcomes will also be compared using treatment-stratified summary statistics, and p-values obtained using the aforementioned statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients >18 who present to the urology clinic at IRL or 3RC with a symptomatic UTI: symptoms include urgency, frequency, urgency urinary incontinence increased from baseline symptoms, dysuria, fevers, flank pain, suprapubic pain/pressure, low back pain, cloudy urine, malodorous urine

Exclusion Criteria:

* patients who are asymptomatic, have an indwelling catheter, SPT, stent, nephrostomy tube, perform CIC, are on daily antibiotic prophylaxis, or already on existing antibiotics

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Contamination | 1 year
  rate of contamination of midstream clean catch urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Joanna A Orzel, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States